CLINICAL TRIAL: NCT03529357
Title: Implementation of Biological Age in Worksite Health Promotion - a Cohort Study on >4000 Danish Employees and Their Health Risk Reductions
Brief Title: Biological Age in Worksite Health Promotion
Acronym: BA1
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Metropolitan University College (Other); Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Jørn Wulff Helge, Ph.D., Proffesor Jørn Wulff Helge, University of Copenhagen
Other Study IDs: BiologicalAge1
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Health Behavior; Biomedical Technology
Keywords: Biological Age; Motivation
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cohort study investigates how implementation of Biological Age technology in worksite health promotion, affects health behavior in the general Danish working population.

DETAILED DESCRIPTION:
This cohort study is designed on the basis of Body Age tests, executed by a private Danish health care company in the period from 2010 to 2013.

The dataset comprises pre- and post Body Age tests from >4000 individuals. They used a standardised protocol and educated staff ( physiotherapists or with a degree in sports science) to carry out the tests. Body Age tests apply biometrics, fitness level and health status data of the employee. The test results are characterized by a Body Age score, which defines the employee's biological age (in years).

This design categorises as a register study why The Danish National Committee is not applied for.

ELIGIBILITY:
Inclusion Criteria:

* Males and females interested in their personal health status
* Participants who perform both baseline and follow up test.

Exclusion Criteria:

* Use of beta blockers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The volunteers are employees in either private or governmental companies. A total of 18 different companies are included in this study, primarily related to banking, pension and pharmaceutical work areas. The Body Age test is voluntary and part of the companies health strategy and fringe benefits.
Sampling Method: Non-Probability Sample
Enrollment: 5473 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Biological Age | The Biological Age is calculated at baseline and at one year follow up
  An algorithm calculates Biological Age, using physiological parameters and biomarkers measured during the test.

SECONDARY OUTCOMES:
BMI | Measured at baseline and at one year follow up
  BodyMassIndex is a major risk factor for developing lifestyle related diseases.
Bodyweight | Measured at baseline and at one year follow up
  The weight in kilograms of each individual
FM | Measured at baseline and at one year follow up
  Fat Mass is important to look at isolated in reference to whole bodyweight
FFM | Measured at baseline and at one year follow up
  Fat Free Mass is important to look at isolated in reference to Whole bodyweight
BP | Measured at baseline and at one year follow up
  Bloodpressure as a result from systolic and diastolic bloodpressure
VO2max | Measured at baseline and at one year follow up
  Maximal Oxygen consumption
BG | Measured at baseline and at one year follow up
  Blood Glucose
HDL | Measured at baseline and at one year follow up
  High Density Lipoprotein
LDL | Measured at baseline and at one year follow up
  Low Density Lipoprotein

CONTACTS AND LOCATIONS:
Overall Officials: Jørn W Helge, Prof., Principal Investigator — BMI, Xlab
Locations (1):
- University of Copenhagen, Department of Biomedical Sciences, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided